CLINICAL TRIAL: NCT01332370
Title: Prescription Patterns, Resource Utilization & Costs - Add-on Therapy With Anti Dipeptidyl Peptidase-IVs vs Rosiglitazone
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112611
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Retrospective; Type 2 Diabetes; Cost Analysis; Rosiglitazone; Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination; Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with Type 2 Diabetes: Subjects with a diagnosis (ICD-9 code) of diabetes
  Interventions: Drug: Rosiglitazone + Metformin; Drug: Sitagliptin + Metformin

INTERVENTIONS:
Drug: Rosiglitazone + Metformin — At least 180 days of continuous therapy with RSG+MET after the first Rx for RSG
  Other Names: Avandia(TM)
Drug: Sitagliptin + Metformin — At least 180 days of continuous therapy with STG+MET after the first Rx for STG
  Other Names: Januvia(R)

SUMMARY:
This retrospective database study analyzed resource utilization and costs associated with sitagliptin (STG) in comparison with rosiglitazone (RSG) added to metformin (MET) monotherapy among adults with a diagnosis of diabetes who were continuously enrolled in a large US healthcare plan.

ELIGIBILITY:
Inclusion Criteria:

* Continuously enrolled in the health insurance plan to ensure complete claims coverage
* At least 1 claim with a diagnosis of diabetes (ICD-9 250.xx)
* Aged 18 years or older at the index date
* At least 6 months of baseline period prior to the index date
* At least 1 claim for MET during the baseline period
* At least 180 days of continuous therapy with RSG+MET or STG+MET after the index date

Exclusion Criteria:

* At least 1 claim for insulin or sulfonylurea in the baseline period
* At least 1 claim with a diagnosis of congestive heart failure in the baseline period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults continuously enrolled in a large US health insurance plan with a diagnosis of diabetes who are currently receiving Metformin
Sampling Method: Non-Probability Sample
Enrollment: 5391 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
medical resource utilization | at least 12 months following first prescription with RSG or STG as an add-on therapy to MET monotherapy.
  Direct healthcare and indirect sick leave costs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline